CLINICAL TRIAL: NCT03786276
Title: Effects of Active Virtual Reality Working Memory Retraining on Heavy Drinking Veterans With Mild Traumatic Brain Injury
Brief Title: Virtual Reality- Working Memory Retraining
Acronym: VR-WMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VR-WMR
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Alcohol Use Disorder; Mild Traumatic Brain Injury
Keywords: Alcohol Use Disorder; Traumatic Brain Injury; Working Memory Training; Virtual Reality; Physical Exercise
MeSH Terms: conditions — Alcoholism; Brain Concussion; Brain Injuries, Traumatic; Motor Activity

STUDY DESIGN:
Intervention Model Description: We will use an 8-week, randomized cross--over design trial of active VR-WMR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise-Only (Experimental): Exercise-Only condition, 12 exercise sessions on a stationary recumbent bicycle over 4 weeks. After 4 weeks, the participants will have a 1-week washout followed by Active VR-WMR arm.
  Interventions: Behavioral: Exercise-only
- VR-WMR-Only (Experimental): Virtual Reality Working Memory Retraining-Only condition, 12 working memory retraining sessions over 4 weeks. After 4 weeks, the participants will have a 1-week washout followed by Active VR-WMR arm.
  Interventions: Behavioral: VR-WMR-Only
- Active VR-WMR (Experimental): After 4 weeks in one of the first two arms, the participants will have a 1-week washout followed by the Active VR-WMR arm. Participants will complete 12 Active VR-WMR sessions on a stationary recumbent bicycle over 4 weeks.
  Interventions: Behavioral: Active VR-WMR

INTERVENTIONS:
Behavioral: VR-WMR-Only — Participants will spend up to 30 minutes in a VR-WMR environment during each training session.
  Other Names: Virtual Reality-Working Memory Retraining
  Arms: VR-WMR-Only
Behavioral: Exercise-only — Participants will ride a stationary recumbent bicycle for up to 30 minutes during each training session.
  Other Names: Recumbent bicycle
  Arms: Exercise-Only
Behavioral: Active VR-WMR — Participants will spend up to 30 minutes in a VR-WMR environment while riding a stationary, recumbent bicycle during each training session.
  Other Names: Active Virtual Reality-Working Memory Retraining
  Arms: Active VR-WMR

SUMMARY:
This study will establish the acceptability and feasibility of enrolling and retaining heavy drinking Veterans with mild traumatic brain injury (mTBI) in an 8-week, randomized cross-over design trial of active VR working memory retraining (WMR). This study will also seek to establish the efficacy of active VR-WMR to increase performance in executive function.

DETAILED DESCRIPTION:
The investigators will employ a physically active VR working memory retraining (VR-WMR) regimen utilizing components of Blue Goji VR Active Gaming. The synthesis of physical activity and an enriched VR environment is expected to yield superior working memory training stemming from greater neurological activation. This enhanced working memory training task will result in greater motivation to engage and complete a training regimen, thus fostering greater improvements in executive function than traditional working memory training tasks; ultimately resulting in increased self-control over alcohol use and other high-risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* must report "heavy" drinking by NIH/NIAAA criteria (>7 drinks/week for women; >14 drinks/week for men) for at least one week in the last 90 days
* must meet moderate to severe criteria for current (past year) alcohol use disorder (AUD) by DSM-5
* must express a desire to reduce, stop, or maintain cessation of alcohol use
* must report a history of TBI as defined by American Congress of Rehabilitation Medicine (ACRM), in the chronic, stable phase of recovery (>6 months from injury)

Exclusion Criteria:

* Unstable medical or psychiatric disorders judged to be unstable in the clinical judgment of the PI
* Current or past history of intrinsic cerebral tumors, HIV infection, cerebrovascular accident, aneurysm, arteriovenous malformations, myocardial infarction, cerebrovascular or peripheral vascular disease, type-1 diabetes, any cardiac, hepatic or renal diseases/disorders, surgical implantation of neurostimulators or cardiac pacemakers, medically diagnosed chronic obstructive pulmonary disease, demyelinating and neurodegenerative diseases, history of seizure disorder, and/or any physical disability making it impossible to use exercise equipment
* No female participant will be pregnant or attempting to conceive
* Concurrent participation in an AUD, cognitive training, or exercise study
* Must not require acute medical detoxification from alcohol (CIWA-AD > 11) within the past week prior to study entry
* Subjects who, in the opinion of the investigator, are otherwise unsuitable for a study of this type will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | 18 months
  A validated measure of technology usability will be administered at end of study to assess the usability of Active VR-WMR.The System Usability Scale (SUS) is a reliable 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree used to measure product usability. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. An SUS score above a 68 would be considered above average and anything below 68 is below average.
The Client Satisfaction Questionnaire | 18 months
  A validated measure of client satisfaction with an intervention will be administered at the end of study to evaluate satisfaction with Active VR-WMR. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction. A standard mean rating of ≥ 24 will be considered acceptable.

SECONDARY OUTCOMES:
Working Memory | 18 months
  Change in working memory in each arm will be evaluated. Working Memory consists of well validated WAIS-IV Arithmetic and Digit Span Subscales. Working memory will be the average of the scaled scores (ss) of each subscale, with a mean (M) = 10 and a standard deviation (SD) = 3. The subtest ss range from 1 to 19.

CONTACTS AND LOCATIONS:
Overall Officials: David L Pennington, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- VA Medical Center San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Pennington DL, Reavis JV, Cano MT, Walker E, Batki SL. The Impact of Exercise and Virtual Reality Executive Function Training on Cognition Among Heavy Drinking Veterans With Traumatic Brain Injury: A Pilot Feasibility Study. Front Behav Neurosci. 2022 Mar 22;16:802711. doi: 10.3389/fnbeh.2022.802711. eCollection 2022. PMID 35391785